CLINICAL TRIAL: NCT05313477
Title: The Effects of Vitamin D and Calcium Supplementation to Parathyroid Hormone in CHB Patients Treated With Tenofovir Disoproxil Fumarate
Brief Title: The Effects of Vitamin D and Calcium Supplementation to Parathyroid Hormone in CHB Patients Treated With TDF
Acronym: TDF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate professor, Faculty of Medicine, Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si 1045/2020
Record Dates: First submitted 2022-03-07; First posted 2022-04-06 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Parathyroid Hormone; Tenofovir Disoproxil Fumarate; Chronic Hepatitis B Virus; Vitamin D
Keywords: Tenofovir disoproxil fumarate; Tenofovir; Chronic hepatitis B; Parathyroid hormone; Bone mineral density; Renal phosphate loss; Vitamin D; Calcium; TDF; PTH; CHB; HBV
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Ergocalciferols; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement group (Active Comparator): Vitamin D2 supplement based on initial vitamin D level
  * ≥ 20ng/mL -> vitamin D2 20,000unit/week
  * 10-19.9ng/mL -> vitamin D2 40,000unit/week
  * <10ng/mL -> vitamin D2 60,000unit/week Calcium carbonate 1000mg/day
  Interventions: Drug: Ergocalciferol Capsules; Drug: Calcium carbonate
- No supplement group (No Intervention): no medication supplement

INTERVENTIONS:
Drug: Ergocalciferol Capsules — Depend on initial 25(OH) vitamin D level If <10ng/mL, 60000U of Ergocalciferol capsules per week If 10-19.9ng/mL, 40000U of Ergocalciferol capsules per week If >20 ng/mL, 20000U of Ergocalciferol capsule per week
  Arms: Supplement group
Drug: Calcium carbonate — 1000mg of Calcium carbonate daily
  Arms: Supplement group

SUMMARY:
Nucleot(s)ide is an antiviral drug that can reduce the number of viruses, reduce the risk of HCC, regress hepatic fibrosis and reduce death from Hepatitis B viral infection. Tenofovir disoproxil fumarate (TDF) is one of nucleotide analogue that is recommended to treated patients with Hepatitis B viral infection. However, long-term TDF therapy may have side effects especially nephrotoxicity and bone toxicity.

Previous studies in human immunodeficiency virus (HIV) infected patients who treated with TDF containing regimen antiretroviral therapy, in vitamin D supplement group had a statistic significance of low parathyroid hormone level and better in bone mineral density regardless of initial vitamin D level. Therefore, the main objective of this study is to evaluate the vitamin D and calcium supplement to patients with hepatitis B who have taken TDF, in parathyroid hormone level, bone mineral density, renal function and renal phosphate loss compared to patients who have no vitamin D and calcium supplement.

DETAILED DESCRIPTION:
Hepatitis B virus is a global public health problem. This infection leads to chronic hepatitis, cirrhosis and liver cancer. According to past statistics, infection with hepatitis B virus is a common cause of hepatocellular carcinoma about 60% in East-Asia and Africa and about 20% in Western countries. About 350-400 million people are infected worldwide. Infection with hepatitis B virus is also an important factor of death in 1million patients per year.

Nucleot(s)ide is an antiviral drug that can reduce the number of viruses, reduce the risk of HCC, regress hepatic fibrosis and reduce death from Hepatitis B viral infection. Nowadays, the recommendation of nucleot(s)ide prefers Tenofovir disoproxil fumarate (TDF), Tenofovir Alafenamide (TAF) and Entecavir (ETV) than Lamivudine, Adefovir and Telbivudine due to high potency and low resistance rate Tenofovir disoproxil fumarate (TDF) is one of nucleotide analogue that inhibits reverse transcriptase in HBV replication process. However, long-term TDF therapy may have side effects especially nephrotoxicity. The proposed mechanisms of nephrotoxicity of TDF are cumulative of TDF at proximal tubule of kidney leads to mitochondrial toxicity, downregulation of sodium-phosphorus cotransporter, sodium/ hydrogen exchanger 3 and aquaporin 2, decreased endothelial nitric oxide-synthase (eNOS) and renal vasoconstriction results in tubulopathy in renal proximal tubule, increase of phosphate loss in urine and increase od serum creatinine.

Moreover, TDF also affects to decrease bone mineral density (BMD) that related with renal phosphate loss, loss of osteoblast function, high parathyroid hormone level regardless of vitamin D level and high fibroblast growth factor 23 (FGF23) leads to worsen in bone mineralization Vitamin D has a protective effect and indicate for osteoporosis treatment. The chronic hepatitis B infected patients with vitamin D deficiency may have a poor prognosis in hepatic fibrosis and high HBV DNA level. Previous studies in human immunodeficiency virus (HIV) infected patients who treated with TDF containing regimen antiretroviral therapy, in vitamin D supplement group had a statistic significance of low parathyroid hormone level and better in bone mineral density regardless of initial vitamin D level. Therefore, the main objective of this study is to evaluate the vitamin D and calcium supplement to patients with hepatitis B who have taken TDF, in parathyroid hormone level, bone mineral density, renal function and renal phosphate loss compared to patients who have no vitamin D and calcium supplement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 75 years old
* Chronic hepatitis B infected patients treated with TDF monotherapy
* eGFR ≥ 60 mL/ min/ 1.73 m2
* HBV viral load <10 IU/ mL

Exclusion Criteria:

* HIV infection or hepatitis C co-infection
* Decompensated cirrhosis, including variceal bleeding, ascites, hepatic encephalopathy
* History of Hepatocellular carcinoma
* Active malignancy of cancer in other organs
* Pregnancy or lactation
* Primary hyperparathyroidism
* History of thyroid or parathyroid surgery
* History of radiation at neck area
* Any osteoporosis treatment or history of osteoporosis diagnosis
* Chronic kidney disease
* Current use of Vitamin D
* Adverse event or allergy to TDF
* Chronic hepatitis B patients with TDF resistance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in serum parathyroid hormone | 48weeks
  Change from the baseline in serum parathyroid hormone as assessed by Electrochemiluminescent immunoassay (ECLIA)

SECONDARY OUTCOMES:
Change in bone mineral density | 48weeks
  Change from the baseline in bone mineral density as assessed by Dual-energy X-ray absorptiometry (DXA)
Renal function changes | 48weeks
  Change from the baseline in renal function (eGFR) based on creatinine as assessed by Enzymatic method
Change in renal phosphate loss | 48weeks
  Change from the baseline in the tubular reabsorption of phosphate (TRP) as renal phosphate loss depended on serum creatinine, urine creatine (assessed by enzymatic method) and serum phosphate, urine phosphate (assessed by modification of the classical phosphomolybdate method by Fiske and Subbarow)

CONTACTS AND LOCATIONS:
Overall Officials: Watcharasak Chotiyaputta, Asso Prof, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trepo C, Chan HL, Lok A. Hepatitis B virus infection. Lancet. 2014 Dec 6;384(9959):2053-63. doi: 10.1016/S0140-6736(14)60220-8. Epub 2014 Jun 18. PMID 24954675
- [Result] Lai CL, Yuen MF. Chronic hepatitis B--new goals, new treatment. N Engl J Med. 2008 Dec 4;359(23):2488-91. doi: 10.1056/NEJMe0808185. No abstract available. PMID 19052131
- [Result] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Result] Zampino R, Boemio A, Sagnelli C, Alessio L, Adinolfi LE, Sagnelli E, Coppola N. Hepatitis B virus burden in developing countries. World J Gastroenterol. 2015 Nov 14;21(42):11941-53. doi: 10.3748/wjg.v21.i42.11941. PMID 26576083
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Result] Yuen MF, Chen DS, Dusheiko GM, Janssen HLA, Lau DTY, Locarnini SA, Peters MG, Lai CL. Hepatitis B virus infection. Nat Rev Dis Primers. 2018 Jun 7;4:18035. doi: 10.1038/nrdp.2018.35. PMID 29877316
- [Result] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Result] Wang YJ, Yang L, Zuo JP. Recent developments in antivirals against hepatitis B virus. Virus Res. 2016 Feb 2;213:205-213. doi: 10.1016/j.virusres.2015.12.014. Epub 2015 Dec 28. PMID 26732483
- [Result] Wong GL, Seto WK, Wong VW, Yuen MF, Chan HL. Review article: long-term safety of oral anti-viral treatment for chronic hepatitis B. Aliment Pharmacol Ther. 2018 Mar;47(6):730-737. doi: 10.1111/apt.14497. Epub 2018 Jan 22. PMID 29359487
- [Result] de Fraga RS, Van Vaisberg V, Mendes LCA, Carrilho FJ, Ono SK. Adverse events of nucleos(t)ide analogues for chronic hepatitis B: a systematic review. J Gastroenterol. 2020 May;55(5):496-514. doi: 10.1007/s00535-020-01680-0. Epub 2020 Mar 17. PMID 32185517
- [Result] Liborio AB, Andrade L, Pereira LV, Sanches TR, Shimizu MH, Seguro AC. Rosiglitazone reverses tenofovir-induced nephrotoxicity. Kidney Int. 2008 Oct;74(7):910-8. doi: 10.1038/ki.2008.252. Epub 2008 Jun 18. PMID 18563054
- [Result] Birkus G, Hitchcock MJ, Cihlar T. Assessment of mitochondrial toxicity in human cells treated with tenofovir: comparison with other nucleoside reverse transcriptase inhibitors. Antimicrob Agents Chemother. 2002 Mar;46(3):716-23. doi: 10.1128/AAC.46.3.716-723.2002. PMID 11850253
- [Result] Kohler JJ, Hosseini SH, Hoying-Brandt A, Green E, Johnson DM, Russ R, Tran D, Raper CM, Santoianni R, Lewis W. Tenofovir renal toxicity targets mitochondria of renal proximal tubules. Lab Invest. 2009 May;89(5):513-9. doi: 10.1038/labinvest.2009.14. Epub 2009 Mar 9. PMID 19274046
- [Result] Rodriguez-Novoa S, Labarga P, Soriano V, Egan D, Albalater M, Morello J, Cuenca L, Gonzalez-Pardo G, Khoo S, Back D, Owen A. Predictors of kidney tubular dysfunction in HIV-infected patients treated with tenofovir: a pharmacogenetic study. Clin Infect Dis. 2009 Jun 1;48(11):e108-16. doi: 10.1086/598507. PMID 19400747
- [Result] Lampertico P, Chan HL, Janssen HL, Strasser SI, Schindler R, Berg T. Review article: long-term safety of nucleoside and nucleotide analogues in HBV-monoinfected patients. Aliment Pharmacol Ther. 2016 Jul;44(1):16-34. doi: 10.1111/apt.13659. Epub 2016 May 19. PMID 27198929
- [Result] Grant PM, Cotter AG. Tenofovir and bone health. Curr Opin HIV AIDS. 2016 May;11(3):326-32. doi: 10.1097/COH.0000000000000248. PMID 26859637
- [Result] Fontana RJ. Side effects of long-term oral antiviral therapy for hepatitis B. Hepatology. 2009 May;49(5 Suppl):S185-95. doi: 10.1002/hep.22885. PMID 19399802
- [Result] Fong TL, Lee BT, Tien A, Chang M, Lim C, Ahn A, Bae HS. Improvement of bone mineral density and markers of proximal renal tubular function in chronic hepatitis B patients switched from tenofovir disoproxil fumarate to tenofovir alafenamide. J Viral Hepat. 2019 May;26(5):561-567. doi: 10.1111/jvh.13053. Epub 2019 Jan 16. PMID 30576085
- [Result] Grigsby IF, Pham L, Mansky LM, Gopalakrishnan R, Carlson AE, Mansky KC. Tenofovir treatment of primary osteoblasts alters gene expression profiles: implications for bone mineral density loss. Biochem Biophys Res Commun. 2010 Mar 26;394(1):48-53. doi: 10.1016/j.bbrc.2010.02.080. Epub 2010 Feb 18. PMID 20171173
- [Result] Masia M, Padilla S, Robledano C, Lopez N, Ramos JM, Gutierrez F. Early changes in parathyroid hormone concentrations in HIV-infected patients initiating antiretroviral therapy with tenofovir. AIDS Res Hum Retroviruses. 2012 Mar;28(3):242-6. doi: 10.1089/AID.2011.0052. Epub 2011 Jul 19. PMID 21639815
- [Result] Mingione A, Maruca K, Chiappori F, Pivari F, Brasacchio C, Quirino T, Merelli I, Soldati L, Bonfanti P, Mora S. High parathyroid hormone concentration in tenofovir-treated patients are due to inhibition of calcium-sensing receptor activity. Biomed Pharmacother. 2018 Jan;97:969-974. doi: 10.1016/j.biopha.2017.11.037. Epub 2017 Nov 7. PMID 29136775
- [Result] Havens PL, Kiser JJ, Stephensen CB, Hazra R, Flynn PM, Wilson CM, Rutledge B, Bethel J, Pan CG, Woodhouse LR, Van Loan MD, Liu N, Lujan-Zilbermann J, Baker A, Kapogiannis BG, Gordon CM, Mulligan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 063 Study Team. Association of higher plasma vitamin D binding protein and lower free calcitriol levels with tenofovir disoproxil fumarate use and plasma and intracellular tenofovir pharmacokinetics: cause of a functional vitamin D deficiency? Antimicrob Agents Chemother. 2013 Nov;57(11):5619-28. doi: 10.1128/AAC.01096-13. Epub 2013 Sep 3. PMID 24002093
- [Result] Childs KE, Fishman SL, Constable C, Gutierrez JA, Wyatt CM, Dieterich DT, Mullen MP, Branch AD. Short communication: Inadequate vitamin D exacerbates parathyroid hormone elevations in tenofovir users. AIDS Res Hum Retroviruses. 2010 Aug;26(8):855-9. doi: 10.1089/aid.2009.0308. PMID 20672993
- [Result] Noe S, Heldwein S, Wiese C, Pascucci R, von Krosigk A, Schabaz F, Jonsson-Oldenbuettel C, Jaeger H, Wolf E. Tenofovir Disoproxil Fumarate Is Associated with a Set-Point Variation in the Calcium-Parathyroid Hormone-Vitamin D Axis: Results from a German Cohort. Adv Pharmacol Sci. 2018 Dec 31;2018:6069131. doi: 10.1155/2018/6069131. eCollection 2018. PMID 30687401
- [Result] Havens PL, Stephensen CB, Hazra R, Flynn PM, Wilson CM, Rutledge B, Bethel J, Pan CG, Woodhouse LR, Van Loan MD, Liu N, Lujan-Zilbermann J, Baker A, Kapogiannis BG, Mulligan K; Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions 063 study team. Vitamin D3 decreases parathyroid hormone in HIV-infected youth being treated with tenofovir: a randomized, placebo-controlled trial. Clin Infect Dis. 2012 Apr;54(7):1013-25. doi: 10.1093/cid/cir968. Epub 2012 Jan 19. PMID 22267714
- [Result] Saeedi R, Mojebi-Mogharar A, Sandhu SK, Dubland JA, Ford JA, Yousefi M, Pudek M, Holmes DT, Erb SR, Peter Kwan W, Kendler DL, Yoshida EM. Lamivudine, Entecavir, or Tenofovir Treatment of Hepatitis B Infection: Effects on Calcium, Phosphate, FGF23 and Indicators of Bone Metabolism. Ann Hepatol. 2017 March-April;16(2):207-214. doi: 10.5604/16652681.1231577. PMID 28233741
- [Result] Havens PL, Hazra R, Stephensen CB, Kiser JJ, Flynn PM, Wilson CM, Rutledge B, Bethel J, Pan CG, Woodhouse LR, Van Loan MD, Liu N, Lujan-Zilbermann J, Baker A, Kapogiannis BG, Gordon CM, Mulligan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 063 study team. Vitamin D3 supplementation increases fibroblast growth factor-23 in HIV-infected youths treated with tenofovir disoproxil fumarate. Antivir Ther. 2014;19(6):613-8. doi: 10.3851/IMP2755. Epub 2014 Feb 17. PMID 24535626
- [Result] Reid IR, Bolland MJ, Grey A. Effects of vitamin D supplements on bone mineral density: a systematic review and meta-analysis. Lancet. 2014 Jan 11;383(9912):146-55. doi: 10.1016/S0140-6736(13)61647-5. Epub 2013 Oct 11. PMID 24119980
- [Result] Reid IR. Vitamin D Effect on Bone Mineral Density and Fractures. Endocrinol Metab Clin North Am. 2017 Dec;46(4):935-945. doi: 10.1016/j.ecl.2017.07.005. Epub 2017 Sep 29. PMID 29080644
- [Result] Hoan NX, Tong HV, Song LH, Meyer CG, Velavan TP. Vitamin D deficiency and hepatitis viruses-associated liver diseases: A literature review. World J Gastroenterol. 2018 Jan 28;24(4):445-460. doi: 10.3748/wjg.v24.i4.445. PMID 29398866
- [Result] Overton ET, Chan ES, Brown TT, Tebas P, McComsey GA, Melbourne KM, Napoli A, Hardin WR, Ribaudo HJ, Yin MT. Vitamin D and Calcium Attenuate Bone Loss With Antiretroviral Therapy Initiation: A Randomized Trial. Ann Intern Med. 2015 Jun 16;162(12):815-24. doi: 10.7326/M14-1409. PMID 26075752
- [Result] Havens PL, Stephensen CB, Van Loan MD, Schuster GU, Woodhouse LR, Flynn PM, Gordon CM, Pan CG, Rutledge B, Harris DR, Price G, Baker A, Meyer WA 3rd, Wilson CM, Hazra R, Kapogiannis BG, Mulligan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 109 Study Team. Vitamin D3 Supplementation Increases Spine Bone Mineral Density in Adolescents and Young Adults With Human Immunodeficiency Virus Infection Being Treated With Tenofovir Disoproxil Fumarate: A Randomized, Placebo-Controlled Trial. Clin Infect Dis. 2018 Jan 6;66(2):220-228. doi: 10.1093/cid/cix753. PMID 29020329